CLINICAL TRIAL: NCT01554696
Title: A Phase 2b, Randomized, Double-blind, Parallel-group, Placebo Controlled, Dose-finding, Multi-center Study to Evaluate the Safety and Efficacy of ASP015K in Moderate to Severe Rheumatoid Arthritis in Patients Who Have Had an Inadequate Response to Methotrexate
Brief Title: A Study to Evaluate the Safety and Efficacy of ASP015K in Moderate to Severe Rheumatoid Arthritis Subjects Who Have Had an Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 015K-CL-RA21; 2011-006018-15 (EudraCT Number)
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Arthritis, Rheumatoid
Keywords: ASP015K; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — peficitinib; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ASP015K lowest dose (Experimental): ASP015K lowest dose daily in addition to concomitant weekly oral methotrexate
  Interventions: Drug: peficitinib; Drug: methotrexate
- ASP015K low dose (Experimental): ASP015K low dose daily in addition to concomitant weekly oral methotrexate
  Interventions: Drug: peficitinib; Drug: methotrexate
- ASP015K medium dose (Experimental): ASP015K medium dose daily in addition to concomitant weekly oral methotrexate
  Interventions: Drug: peficitinib; Drug: methotrexate
- ASP015K high dose (Experimental): ASP015K high dose daily in addition to concomitant weekly oral methotrexate
  Interventions: Drug: peficitinib; Drug: methotrexate
- Placebo (Placebo Comparator): Placebo daily in addition to concomitant weekly oral methotrexate
  Interventions: Drug: Placebo; Drug: methotrexate

INTERVENTIONS:
Drug: peficitinib — oral
  Other Names: ASP015K
  Arms: ASP015K high dose; ASP015K low dose; ASP015K lowest dose; ASP015K medium dose
Drug: Placebo — oral
  Arms: Placebo
Drug: methotrexate — oral

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of ASP015K in moderate to severe rheumatoid arthritis subjects who are methotrexate-inadequate responders (MTX-IR).

DETAILED DESCRIPTION:
Subjects in each treatment group will continue to take their concomitant oral weekly dose of methotrexate (MTX) in addition to daily ASP015K or matching placebo, taken orally with food, daily for 12 weeks after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Subject has rheumatoid arthritis (RA) diagnosed according to the 1987 revised ACR criteria for at least 6 months prior to Screening
* Subject has been treated with oral methotrexate (MTX) for a minimum of 90 days and at a stable dose for 28 days prior to the first dose of study drug
* ≥6 tender/painful joints; ≥6 swollen joints
* Subject meets the ACR 1991 Revised Criteria for Global Functional Status in RA Class I, II or III at Screening and Baseline
* Subject's other medication taken for treatment of RA must be stable for at least 28 days prior to start of the study
* Male and female subjects must be willing to comply with contraception requirements as well as restrictions regarding egg and sperm donation
* Female subject must not be breastfeeding at Screening or during the study period, and for 60 days after the final study drug administration
* Subject agrees not to participate in another interventional study while on treatment

Exclusion Criteria:

* Positive Mycobacterium tuberculosis (TB) test within 90 days of Screening
* Abnormal chest x-ray indicative of an acute or chronic infectious process or malignancy
* Receipt of live or live attenuated virus vaccination within 30 days prior to the first dose of study drug
* Known history of positive test for hepatitis B surface antigen (HBsAg) or hepatitis C antibody or history of a positive test for human immunodeficiency virus (HIV) infection
* History of any other autoimmune rheumatic disease, other than Sjogren's syndrome
* Previous history of clinically significant infections or illness (requiring hospitalization or requiring parenteral therapy) within 90 days of the Baseline visit, or a history of any illness that would preclude participation in the study
* History of any malignancy, except for successfully treated basal or squamous cell carcinoma of the skin or in-situ carcinoma of the cervix
* Does not meet specified washout criteria for the following RA medications: gold, azathioprine, minocycline, penicillamine, etanercept, certolizumab, adalimumab, golimumab, infliximab, cyclophosphamide, and leflunomide
* Subject has previously used a non anti-TNF biologic disease-modifying antirheumatic drug (DMARD) (e.g., anakinra, abatacept, rituximab, tocilizumab)
* Previous intolerance to Janus kinase (JAK) inhibitors
* Receipt of intra-articular or parenteral corticosteroid within 28 days prior to the first dose of study drug or is currently taking > 30 mg oral morphine (or narcotic equivalent) per day
* Absolute lymphocyte count (ALC) < 750/mm3
* Receipt of plasma exchange therapy within 60 days prior to the start of study drug
* Receipt of any investigational agent within 30 days or 5 half-lives, whichever is longer, prior to first dose of study drug
* Receipt of medications that are CYP3A substrates with narrow therapeutic range within 14 days prior to first dose of study drug
* History of heart failure, defined as New York Heart Association (NYHA) grade 3 or greater
* History of long QT syndrome or prolonged QT interval
* Any ongoing severe, progressive, or uncontrolled renal, hepatic, hematological, gastrointestinal, metabolic, endocrine, pulmonary, cardiac, neurological, or infectious disease, or any ongoing illness which would make the subject unsuitable for the study. This includes stomatitis, gastrointestinal ulcers, or any other condition that would preclude continued treatment with methotrexate
* Subject has any condition possibly affecting oral absorption (e.g., gastrectomy, other malabsorption syndromes, or clinically significant diabetic gastroenteropathy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 379 (Actual)
Dates: Start 2012-07-06 (Actual); Primary Completion 2014-02-11 (Actual); Study Completion 2014-02-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects achieving American College of Rheumatology Criteria 20 (ACR 20) response | Week 12
Trough plasma concentration of ASP015K and metabolite(s) | up to Week 12

SECONDARY OUTCOMES:
Percentage of subjects achieving ACR 50 response | Week 12
Percentage of subjects achieving ACR 70 response | Week 12
Change from baseline in Disease Activity Score using 28 joint count and C Reactive Protein (DAS28-CRP) | Baseline and Week 12

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director Director, Study Director — Astellas Pharma Global Development
Locations (49):
- United States (19):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - The Talbert Group, Huntington Beach, California
  - University of California San Diego, La Jolla, California
  - Desert Medical Advances, Palm Desert, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Arthritis Associates of Colorado Springs, Colorado Springs, Colorado
  - Arthritis Associates, Orlando, Florida
  - Illinois Bone & Joint, Morton Grove, Illinois
  - Deerbrook Medical Asssociates, Vernon Hills, Illinois
  - Center for Arthritis and Osteoporosis, Elizabethtown, Kentucky
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - PMG Research, Hickory, North Carolina
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Clincal Research Center of Reading, Wyomissing, Pennsylvania
  - Rheumatology Consultants, PLLC, Knoxville, Tennessee
  - Austin Rheumatology Research PA, Austin, Texas
  - Center for Arthritis & Rheumatic Disease, P.C., Chesapeake, Virginia
  - Mountain State Clinical Research, Clarksburg, West Virginia
- Belgium (2):
  - Hospital Erasme, Brussels
  - Moliere Hospital, Brussels
- Bulgaria (3):
  - MHAT Burgas, Burgas
  - MHAT Plovdiv AD, Plovdiv
  - MHAT "Sv. Ivan Rilski", Sofia
- Colombia (6):
  - IPS Rodrigo Botero SAS, Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe S.A.S, Barranquilla
  - Centro Integral De Reumatologia E Inmunologia, Bogotá
  - Medicity Sas, Bucaramanga
  - Servimed E.U., Bucaramanga
  - Centro de medicina Interna Julian Coronel, Cali
- Czechia (3):
  - Revmatologicky ustav, Prague
  - MEDICAL PLUS, s.r.o. or REVMACENTRUM UH, s.r.o., Uherské Hradiště
  - PV-MEDICAL s.r.o., Zlín
- Hungary (4):
  - DRC Gyogyszervizsgalo Kozpont Kft, Balatonfüred
  - Rethy Pal Korhaz es Rendelointezet, Békéscsaba
  - Revita Clinic Rheumatology, Budapest
  - Kenezy Hospital Institute of Clinical Pharmacology, Debrecen
- Mexico (5):
  - Morales Vargas Centro de Investigacion, SC Rheumatology, León, Guanajuato
  - Hospital Civil de Guadalajara Fray Antonio Alcalde Gutierrez, Guadalajara
  - Dr Javier Orozco Alcala Private Doctor´s office, Guadalajara
  - Cliditer S.A. de C.V.Huerta S.I., Mexico City
  - Centro de Investigacion Clinica de Morelia, S.C., Morelia
- Poland (7):
  - NZOZ Osteo-Medic sc A. Racewicz, J. Supronik, Bialystok
  - Centrum Osteoporozy i Chorob KKostno-Stawowych Daniluk Clinical Research Centre, Bialystok
  - Szpital Uniwersytecki nr. 2 im. Dr. Jana Biziela, Bydgoszcz
  - NZOZ Centrum Medyczne ProMiMed, Krakow
  - Zespol Poradni Specjalistycznych REUMED sp. Zo.o, Lublin
  - ARS Rheumatica, Warsaw
  - Rheuma Medicus Zaktad Opieki Zdrowotnej Relle Brkolozka, Wraszawa

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Kivitz AJ, Gutierrez-Urena SR, Poiley J, Genovese MC, Kristy R, Shay K, Wang X, Garg JP, Zubrzycka-Sienkiewicz A. Peficitinib, a JAK Inhibitor, in the Treatment of Moderate-to-Severe Rheumatoid Arthritis in Patients With an Inadequate Response to Methotrexate. Arthritis Rheumatol. 2017 Apr;69(4):709-719. doi: 10.1002/art.39955. PMID 27748083
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=322